CLINICAL TRIAL: NCT03763370
Title: Managed Access Program for Belantamab Mafodotin in Combination With Either Bortezomib/Dexamethasone or Pomalidomide/Dexamethasone in Patients With Multiple Myeloma Previously Treated With at Least 1 Prior Line of Therapy
Brief Title: Managed Access Program for Combination Treatment With Belantamab Mafodotin in Multiple Myeloma
Status: Available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 209233
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: 213304; belantamab mafodotin; Bortezomib; Dexamethasone; Pomalidomide; Expanded Access Program; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Belantamab mafodotin 2.5 mg/kg IV Q3Weeks + Vd (BVd) — Drug: Belantamab mafodotin
  •Belantamab mafodotin 2.5 milligram per kilogram (mg/kg) intravenous (IV) will be administered at every cycle, once every 3 Weeks, on Day 1 of every cycle, until completion of treatment.
  Drug: Bortezomib •Bortezomib will be administered based on the full prescribing information, for the first 8 Cycles
  Drug: Dexamethasone
  •Dexamethasone will be administered based on the full prescribing information, for the first 8 Cycles
Drug: Belantamab mafodotin 2.5/1.9 mg/kg IV Q4Weeks + Pd (BPd) — Drug: Belantamab mafodotin:
  * Cycle 1: Belantamab mafodotin 2.5 mg/kg IV administered once
  * Cycle 2 onward: Belantamab mafodotin 1.9 mg/kg IV administered once every 4 weeks until completion of treatment
  Drug: Pomalidomide •Pomalidomide will be administered at every cycle, based on the full prescribing information
  Drug: Dexamethasone
  •Dexamethasone will be administered at every cycle, based on the full prescribing information

SUMMARY:
Compassionate use access to belantamab mafodotin (GSK2857916) (in combination with bortezomib/dexamethasone or pomalidomide/dexamethasone) for eligible participants with multiple myeloma previously treated with at least 1 prior line of therapy.

DETAILED DESCRIPTION:
Belantamab mafodotin (GSK2857916) is an antibody-drug conjugate (ADC) comprised of an afucosylated, humanized Immunoglobulin G1 (IgG1) monoclonal immunoconjugate that binds specifically to B-Cell Maturation Antigen. This program is intended to provide access to belantamab mafodotin (in combination with bortezomib/dexamethasone or pomalidomide/dexamethasone) in patients with Multiple Myeloma (MM) who have received at least 1 prior therapy for multiple myeloma, and whose treating physicians have determined that there is unmet treatment need.

ELIGIBILITY:
Specific eligibility criteria must be met, these include:

1. There is no satisfactory alternative treatment for the patient including approved standard of care treatments for their multiple myeloma; and
2. There is reason to believe that the benefit to the patient using belantamab mafodotin outweighs the risk
3. Patient does not qualify for, or is unable to participate in, other ongoing clinical trials

INCLUSION CRITERIA:

1. Written informed consent
2. Diagnosis of multiple myeloma and/or plasma cell dyscrasias and either:

   1. For combination with bortezomib/dexamethasone; previously treated with at least 1 prior line of MM therapy and must have documented disease progression during or after their most recent therapy OR
   2. For combination with pomalidomide/dexamethasone; have been previously treated with at least 1 prior line of MM therapy including a lenalidomide-containing regimen (lenalidomide must have been administered for at least 2 consecutive cycles) and must have documented disease progression during or after their most recent therapy.
3. Able to obtain ophthalmic examinations at baseline, before the next 3 subsequent treatment cycles and as clinically indicated on treatment
4. Contraception requirements

A. Female Participants: A female patient is eligible to participate if one of the following conditions applies:

I. The patient Is not a woman of childbearing potential (WOCBP) OR II. The patient Is a WOCBP and using an effective contraceptive method during treatment with belantamab mafodotin and for 4 months after the last dose. The patient must also have a negative highly sensitive serum pregnancy test within 72 hours of dosing on Cycle 1 Day 1. Please discuss with GSK physician if the patient is pregnant, breast-feeding or planning to have a baby.

B. Male participants with female partners of child-bearing potential are eligible to participate if they agree to use effective contraception during treatment with belantamab mafodotin until 6 months after the last dose

EXCLUSION CRITERIA:

1. If considering combination with bortezomib/dexamethasone intolerant or refractory to bortezomib. If considering combination with pomalidomide/dexamethasone intolerant or refractory to pomalidomide
2. Alanine transaminase (ALT) >2.5x upper limit of normal (ULN).
3. Total bilirubin >1.5xULN; patients with Gilbert's syndrome can be included with total bilirubin >1.5xULN as long as direct bilirubin is ≤1.5xULN.
4. Cirrhosis or current unstable liver or biliary disease per physician assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, persistent jaundice.
5. Patients with Hepatitis B will be excluded unless:

   1. HbcAb positive, HBsAg negative: HBV deoxyribonucleic acid (DNA) undetectable and Antiviral treatment instituted if HBV DNA becomes detectable
   2. HBsAg positive at screen or within 3 months prior to first dose: HBV DNA undetectable and Antiviral treatment maintained throughout program treatment
6. Patients with positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of program treatment unless:

   1. RNA test negative
   2. Successful anti-viral treatment followed by a negative HCV RNA test after a washout period of at least 4 weeks
7. Evidence of Active Bleeding requiring intervention
8. Currently Active Graft-versus-host disease (GvHD)
9. Known Hypersensitivity to the active substance or to any of the excipients
10. Previous progression on belantamab mafodotin
11. Active infection requiring treatment
12. Previous participation in DREAMM-7 or DREAMM-8 clinical trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: If you are a Healthcare Professional who would like to request compassionate use of a GSK investigational medicine for a patient, please use the GSK Compassionate Use Request Portal. — http://gsk-cu-portal.idea-point.com